CLINICAL TRIAL: NCT00358033
Title: Effectiveness of Different Strategies in Maintaining Target Goals of Cardiovascular Risk Factors in Patients Discharged From Cardiovascular Risk Reduction Clinic
Brief Title: Strategies to Maintain Cardiac Risk Control After Discharge From Cardiovascular Risk Reduction Clinic
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Providence VA Medical Center (U.S. Federal Agency)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Wen-Chih Wu, Staff Cardiologist, Providence VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12712
Record Dates: First submitted 2006-07-24; First posted 2006-07-28 (Estimated); Last update posted 2014-04-16 (Estimated); Status verified 2014-04

CONDITIONS: Diabetes; Dyslipidemia; Hypertension; Coronary Atherosclerosis
MeSH Terms: conditions — Diabetes Mellitus; Dyslipidemias; Hypertension; Coronary Artery Disease | interventions — Counseling; Self-Help Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- group intervention (Experimental): pharmacist-led group intervention in behavioral and pharmacologic therapy
  Interventions: Behavioral: Counseling; Behavioral: Interactive Education; Behavioral: Group Support; Procedure: Pharmacologic case management
- individual (Active Comparator): pharmacist-based individual clinic visits with behavioral and pharmacologic intervention for cardiac risk reduction
  Interventions: Behavioral: Counseling; Procedure: Pharmacologic case management
- usual care (No Intervention): usual care

INTERVENTIONS:
Behavioral: Counseling
  Arms: group intervention; individual
Behavioral: Interactive Education
  Arms: group intervention
Behavioral: Group Support
  Arms: group intervention
Procedure: Pharmacologic case management — Provided by clinical pharmacists
  Arms: group intervention; individual

SUMMARY:
The purpose of this study is to determine whether a combined behavioral and pharmacological intervention provided by a multidisciplinary team will further reduce LDL-C, smoking, BP and Hb-A1C in diabetic patients with A1c between 7% and 9% when compared to usual care.

ELIGIBILITY:
Inclusion Criteria:

* Previous enrollment in Cardiovascular Risk Reduction Clinic (CRRC)
* Eligible for CRRC discharge:

  1. For DM patients:

     * HbA1c < 7.0 %,
     * BP < 130/85 mm Hg , and
     * LDL < 100 mg/dl;
  2. For Non-DM patients:

     * BP < 140/90 mm Hg, and
     * LDL < 100 mg/dl;
* Able and willing to sign informed consent.

Exclusion Criteria:

* Presence of conditions that might limit long-term compliance (eg, dementia, acute psychiatric decompensation within the previous 6 months, unstable psychiatric disorder);
* Metastatic disease or terminal illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2003-07; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
The number of patients who had non-compliance to ADA target goals in smoking, LDL cholesterol, blood pressure or Hb A1c. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Chih Wu, MD, Principal Investigator — Providence VAMC
Locations (1):
- Providence VAMC, Providence, Rhode Island, United States